CLINICAL TRIAL: NCT01201759
Title: Effects of Salsalate on Prandial-Induced Vascular Inflammation After SCI
Brief Title: Effects of Salsalate on Prandial-Induced Vascular Inflammation After Spinal Cord Injury (SCI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Mark S. Nash, Ph.D., FACSM, Professor, University of Miami
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 20090361; TMP-MN-004 (Other: Clinicaltrials.gov)
Record Dates: First submitted 2010-09-08; First posted 2010-09-15 (Estimated); Results first posted 2015-06-10 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: Spinal Cord Injury
Keywords: cardiovascular risk
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo to Salsalate 2gr BID (Experimental): Placebo twice a day for 30 days. Then Salsalate 2gr BID for 30 days.
  Interventions: Drug: Salsalate 2grams twice a day for 30 days. Then Placebo for 30 days; Drug: Placebo twice a day for 30 days. Then Salsalate 2gr BID for 30 days.
- Salsalate 2gr BID to placebo (Experimental): Salsalate 2grams twice a day for 30 days. Then Placebo for 30 days.
  Interventions: Drug: Salsalate 2grams twice a day for 30 days. Then Placebo for 30 days; Drug: Placebo twice a day for 30 days. Then Salsalate 2gr BID for 30 days.

INTERVENTIONS:
Drug: Salsalate 2grams twice a day for 30 days. Then Placebo for 30 days — Participants will undergo randomization to either 1 month of Salsalate (4.0 g/day) or placebo. An untreated wash-in (1 month) will precede treatment (1 month), and a washout cross-over period (1 month) will follow. After the wash-in month participants will receive either Salsalate or the placebo. The last month will test effects of drug-placebo not examined in month 2
Drug: Placebo twice a day for 30 days. Then Salsalate 2gr BID for 30 days. — Participants will undergo randomization to either 1 month of Salsalate (4.0 g/day) or placebo. An untreated wash-in (1 month) will precede treatment (1 month), and a washout cross-over period (1 month) will follow. After the wash-in month participants will receive either Salsalate or the placebo. The last month will test effects of drug-placebo not examined in month 2.

SUMMARY:
The overall study objectives are to examine whether:

1. Persons with spinal cord injury (SCI) having elevated body mass are at greater cardiovascular disease (CVD) risk for fasting and postprandial lipidemia, glycemia, and vascular inflammation than persons with SCI having 'normal' body mass, and
2. An inexpensive, low-risk, widely-available pharmacotherapy safely reduces CVD risks associated with fasting and postprandial lipidemia, glycemia, and vascular inflammation.

DETAILED DESCRIPTION:
To test Study Objective 1, 'overweight' and 'non-overweight' persons with SCI will be compared at baseline for fasting and postprandial responses. For Study Objective 2, all persons tested for Study Objective 1 will undergo randomization to either 1 month of Salsalate (4.0 g/day) or placebo. An untreated wash-in (1 month) will precede treatment (1 month), and a washout cross-over period (1 month) will follow. The last month will test effects of drug-placebo not examined in month 2. Fasting and postprandial responses will be tested at each time point. Intention-to-treat clinical standards ("…as randomized, so analyzed…") and 'last observation carried forward' clinical methods will be adopted.

Participants with tetraplegia are sought, as they have fewer exercise options than those with paraplegia and are at greater risk for sedentary lifestyle resulting in CVD, CVD risks, and obesity.

ELIGIBILITY:
Inclusion Criteria:

* SCI resulting in tetraplegia at C3-C7
* injury for more than one year

Exclusion Criteria:

* 1. any recent dietary or other lifestyle changes;
* 2. diabetes or inflammatory medical conditions;
* 3. a pressure ulcer;
* 4. lung or bladder infection;
* 5. undiagnosed illness or fever;
* 6. recent surgery;
* 7. stomach ulcer or a history of stomach upset when taking aspirin or medicines like aspirin, or ,
* 8. currently taking medicines used for pain or inflammation (aspirin and non-steroidal anti-inflammatory drugs, corticosteroids), blood vessel diseases (statins or fibric acid derivatives), blood clotting disorders (Coumadin, Plavix), infections (antibiotics), diabetes (Metformin), and burning 'central' pain (voltage regulators).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-07; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Nash, PhD, Principal Investigator — University of Miami Miller School of Medicine, The Miami Project to Cure Paralysis
Locations (1):
- The Miami Project to Cure Paralysis, Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants underwent randomization to either 1 month of Salsalate ( 4.0 grams daily in split doses) or placebo.
Pre-assignment Details: An untreated wash-in (1 month) preceded treatment (1 month).A 1 month wash-out between cross-over.
Groups:
- Salsalate to Placebo 2gr BID: Salsalate 2grams twice a day for 30 days. Then Placebo for 30 days.
  Salsalate 2grams twice a day for 30 days. Then Placebo for 30 days: Participants will undergo randomization to either 1 month of Salsalate (4.0 g/day) or placebo. An untreated wash-in (1 month) will precede treatment (1 month), and a washout cross-over period (1 month) will follow. After the wash-in month participants will receive either Salsalate or the placebo. The last month will test effects of drug-placebo not examined in month 2
Period: Visit 1 Wash-in ( Untreated)
Arm/Group | Placebo to Salsalate 2gr BID | Salsalate to Placebo 2gr BID
Started | 10 | 8
Completed | 8 | 7
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 1
Period: Visit 2
Arm/Group | Placebo to Salsalate 2gr BID | Salsalate to Placebo 2gr BID
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0
Period: Visit 3 - Washout
Arm/Group | Placebo to Salsalate 2gr BID | Salsalate to Placebo 2gr BID
Started | 8 | 7
Completed | 7 | 4
Not Completed | 1 | 3
Not completed — Adverse Event | 0 | 3
Not completed — Lost to Follow-up | 1 | 0
Period: Visit 4 Crossover
Arm/Group | Placebo to Salsalate 2gr BID | Salsalate to Placebo 2gr BID
Started | 7 | 4
Completed | 7 | 3
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Period: Visit 5
Arm/Group | Placebo to Salsalate 2gr BID | Salsalate to Placebo 2gr BID
Started | 7 | 3
Completed | 7 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo to Salsalate 2gr BID | Salsalate to Placebo 2gr BID | Total
Number analyzed (Participants) | 10 | 8 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 8 | 18
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (10) | 25 (3) | 33 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 10 | 8 | 18

OUTCOME MEASURES:

1. Primary Outcome: Change in Area Under the Curve (AUC) for Lipemia (Triglycerides) at Visits 2-3 or 4-5 Depending on Order of Treatment Assignment.
Description: The postprandial lipemia is assessed by the change in the AUC for plasma triglycerides sampled before and after intervention at time points 0 (immediately post-feeding)to 480 min.
  For peak TG, and TG area under the curve (AUC), treatments (placebo and salsalate) and visits (pre and post treatment) were defined as within-subject's factors.
Time Frame: Each visit samples at 0 (immediately post-feeding), and 30,60,90,120,240,360,480 min post-feeding..
Population: All enrolled participants who completed the study.
Measure: Mean (Standard Deviation); unit: mg*min/dL
Groups:
- Placebo: Placebo 2 grams twice a day for 30 days. Participants will undergo randomization to either 1 month of Salsalate (4.0 g/day) or placebo. An untreated wash-in (1 month) will precede treatment (1 month), and a washout cross-over period (1 month) will follow. After the wash-in month participants will receive either Salsalate or the placebo. The last month will test effects of drug-placebo not examined in month 2.
- Salsalate: Drug: Salsalate 2grams twice a day for 30 days. Then Placebo for 30 days Participants will undergo randomization to either 1 month of Salsalate (4.0 g/day) or placebo. An untreated wash-in (1 month) will precede treatment (1 month), and a washout cross-over period (1 month) will follow. After the wash-in month participants will receive either Salsalate or the placebo. The last month will test effects of drug-placebo not examined in month 2
Arm/Group | Placebo | Salsalate
Number analyzed (Participants) | 10 | 10
mg*min/dL | -34 (104) | -62 (136)

2. Secondary Outcome: Change in Area Under the Curve (AUC) for Glycemia (Glucose) at Visits 2-3 or 4-5 Depending on Order of Treatment Assignment.
Description: The postprandial glycemia is assessed by the change in the AUC for plasma glucose sampled before and after intervention at time points of 0 (immediately post-feeding) to 480 min.
  For peak Glucose, and Glucose area under the curve (AUC), treatments (placebo and salsalate) and visits (pre and post treatment) were defined as within-subject's factors.
Time Frame: Blood samples for each visit were sampled at 0 (immediately post-feeding), and 30,60,90,120,240,360,480 min post-feeding..
Population: All participants who completed treatment.
Measure: Mean (Standard Deviation); unit: mg*min/dL
Arm/Group | Placebo | Salsalate
Number analyzed (Participants) | 10 | 10
mg*min/dL | 1 (15) | -8 (20)

3. Secondary Outcome: Change in Area Under the Curve (AUC) for Lipemia (Free Fatty Acids ) at Visits 2-3 or 4-5 Depending on Order of Treatment Assignment.
Description: The postprandial lipemia is assessed by the change in the AUC for plasma Free fatty acids (FFA)sampled before and after intervention at time points of 0min immediately post feeding to 480 min.
  For peak FFA area under the curve (AUC), treatments (placebo and salsalate) and visits (pre and post treatment) were defined as within-subject's factors.
Time Frame: Each visit sampled at 0 (immediately post-feeding), and 30,60,90,120,240,360,480 min post-feeding..
Population: All enrolled participants who completed the study.
Measure: Mean (Standard Deviation); unit: mg*min/dL
Groups:
- Placebo: Placebo twice a day for 30 days. Then Salsalate 2gr BID for 30 days.: Participants will undergo randomization to either 1 month of Salsalate (4.0 g/day) or placebo. An untreated wash-in (1 month) will precede treatment (1 month), and a washout cross-over period (1 month) will follow. After the wash-in month participants will receive either Salsalate or the placebo. The last month will test effects of drug-placebo not examined in month 2.
- Salsalate: Salsalate 2grams twice a day for 30 days. Then Placebo for 30 days: Participants will undergo randomization to either 1 month of Salsalate (4.0 g/day) or placebo. An untreated wash-in (1 month) will precede treatment (1 month), and a washout cross-over period (1 month) will follow. After the wash-in month participants will receive either Salsalate or the placebo. The last month will test effects of drug-placebo not examined in month 2
Arm/Group | Placebo | Salsalate
Number analyzed (Participants) | 10 | 10
mg*min/dL | 8 (193) | -111 (174)

4. Secondary Outcome: Change in Fasting Values for Vascular Inflammation IL-6 at Visits 2-3 or 4-5
Description: The pro-atherogenic inflammatory mediators are assessed by the change in fasting values of Interleukin-6 in plasma concentration Pre and Post intervention at -30 min ( fasting).
  For fasting values treatments (placebo and salsalate) and visits (pre and post) were defined as within subject's factors.
Time Frame: Study visit at min -30 (fasting)
Population: All enrolled participants who completed the study.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Salsalate
Number analyzed (Participants) | 10 | 10
mg/dL
  Pre-Intervention | 0.48 (0.35) | 0.51 (0.55)
  Post-Intervention | 0.50 (0.49) | 0.19 (0.53)

ADVERSE EVENTS:
Time Frame: Intervention period (30 days Placebo/Salsalate) .
Description: Population included all participants who received at least one dose of the intervention Placebo or Salsalate.
Groups:
- Placebo 2gr BID: Placebo twice a day for 30 days.
- Salsalate 2gr BID: Salsalate 2grams twice a day for 30 days.
Arm/Group | Placebo 2gr BID | Salsalate 2gr BID
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 3/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo 2gr BID (N=18) | Salsalate 2gr BID (N=18)
Fatigue (General disorders) | 0 (0) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Abdominal Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No